CLINICAL TRIAL: NCT02610400
Title: Targeted Parasite Elimination in the Human and Mosquito to Reduce Malaria Transmission: A Cluster Randomised Controlled Factorial Design Trial of Reactive Focal Drug Administration (rfMDA) Versus Reactive Case Detection (RACD), With and Without Reactive Vector Control (RAVC), From the Low Endemic Setting of Namibia
Brief Title: Evaluation of Reactive Focal Mass Drug Administration (rfMDA) +/- Reactive Focal Vector Control (RAVC) in Namibia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Texas (Other); London School of Hygiene and Tropical Medicine (Other); University of Southampton (Other); The Novartis Foundation (Other); Clinton Health Access Initiative, Nigeria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: OPP1089413_Namibia_rfMDA
Record Dates: First submitted 2015-09-18; First posted 2015-11-20 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- RACD without RAVC (Experimental): In this arm, subjects will receive RACD without the addition of RAVC.
  Interventions: Combination Product: RACD
- RACD+RAVC (Experimental): In this arm, subjects will receive both:
  (i) reactive case detection (RACD) and (ii) additional reactive vector control (RAVC)
  Interventions: Combination Product: RACD; Combination Product: RAVC
- rfMDA without RAVC (Experimental): In this arm, subjects will receive reactive focal mass drug administration (rfMDA) without the addition of RAVC.
  Interventions: Combination Product: RAVC; Combination Product: rfMDA
- rfMDA+RAVC (Experimental): In this arm, subjects will receive both:
  (i) reactive focal mass drug administration (rfMDA) and (ii) RAVC.
  Interventions: Combination Product: rfMDA

INTERVENTIONS:
Combination Product: RACD — Active malaria surveillance using rapid diagnostic test in households around passively-detected index case. RDT-positive subjects are treated per national policy, under which combination medication artemether-lumefantrine is first-line, using dosing (mg artemether / mg lumefantrine):
  (i) 5-14kg patient: 20/120mg twice (8 hr apart) on day 1, 20/120mg twice (12 hr apart) on each of days 2 and 3 then stop (ii) 15-24kg patient: 40/240mg twice (8 hrs apart) on day 1, 40/240mg twice (12 hrs apart) on each of days 2 and 3 then stop (iii) 25-34kg patient: 60/360mg twice (8 hrs apart) on day 1, 60/360mg twice (12 hrs apart) on each of days 2 and 3 then stop (iv) > 34kg patient: 80/480mg twice (8 hrs apart) on day 1, 80/480mg twice (12 hrs apart) on each of days 2 and 3, then stop
  Other Names: Reactive Case Detection
  Arms: RACD without RAVC; RACD+RAVC
Combination Product: RAVC — Focal, targeted indoor spraying with long-lasting insecticide pirimiphos-methyl or Actellic 300 CS, a World Health Organization (WHO)-approved organophosphate. Safety measures: (i) seeking advance permission to spray; (ii) temporarily removing items (utensils, water, food, pets) from the building during spray; (iii) covering all unremovable items; (iv) asking inhabitants to temporarily relocate outdoors during spray; (v) advising children remain outdoors until floors washed; and (vi) avoiding of spraying of any rooms that contain inhabitants, animals, or incorrectly removed/covered items. Actellic will be applied according to National Vector-borne Disease Control Program (NVDCP) indoor residual spraying (IRS) guidelines, using a Hudson X-pert sprayer (Hudson Manufacturing Co., Chicago, USA) at 40 mL/m-sq.
  Other Names: Reactive Vector Control
  Arms: RACD+RAVC; rfMDA without RAVC
Combination Product: rfMDA — Presumptive treatment, using the medication A-L, of the inhabitants of households surrounding a passively-detected index case, without incorporating a diagnostic test step. The investigators will administer A-L with dosing as follows (mg artemether / mg lumefantrine):
  (i) 5-14kg patient: 20/120mg twice (8 hours apart) on day 1, 20/120mg twice (12 hours apart) on each of days 2 and 3, then stop (ii) 15-24kg patient: 40/240mg twice (8 hours apart) on day 1, 40/240mg twice (12 hours apart) on each of days 2 and 3, then stop (iii) 25-34kg patient: 60/360mg twice (8 hours apart) on day 1, 60/360mg twice (12 hours apart) on each of days 2 and 3, then stop (iv) > 34kg patient: 80/480mg twice (8 hours apart) on day 1, 80/480mg twice (12 hours apart) on each of days 2 and 3, then stop
  Other Names: Reactive focal mass drug administration
  Arms: rfMDA without RAVC; rfMDA+RAVC

SUMMARY:
This is a cluster randomised controlled trial with factorial study design comparing the impact of reactive community-based malaria interventions: 1) presumptive treatment (or rfMDA, reactive focal mass drug administration) versus reactive case detection (RACD), and 2) reactive IRS (indoor residual spraying) versus control on the incidence of malaria in Namibia.

DETAILED DESCRIPTION:
In recent years, many countries, including Namibia, have experienced reductions in malaria transmission in association with the scale-up of effective interventions and are now moving towards malaria elimination. In malaria control, the goal is to reduce the clinical burden of malaria. In malaria elimination, the aim is to interrupt transmission, and it becomes necessary to address not only symptomatic malaria, but also asymptomatic infections that contribute to transmission. Since malaria transmission is highly geographically heterogeneous, elimination activities should target hot spots, or areas where the risk of future infection is highest. Hence, in the transition from control to elimination, enhanced surveillance and response is necessary to target hot spots with interventions to interrupt transmission.

Reactive case detection (RACD), active surveillance in communities around passively detected cases, is a recommended elimination strategy to identify secondary cases and hot spots. However, RACD can be labour-, time-, and cost- intensive, and misses people who are absent during screening or refuse to have their blood drawn. Furthermore, both microscopy and rapid diagnostic tests (RDTs) utilized in RACD have shortcomings, for instance, the suboptimal sensitivity of RDTs for low parasite density and non-falciparum infections. Polymerase chain reaction (PCR) offers markedly improved sensitivity over RDTs but requires hours of processing time, sophisticated technical skills, and expensive equipment. Given these limitations, presumptive treatment may be a more feasible and effective strategy to reduce and interrupt transmission.

Reactive focal mass drug administration (rfMDA), a form of presumptive treatment, has been used successfully in China to overcome some of the weaknesses of RACD. rfMDA targets remaining reservoirs of infection in low endemic settings by treating everyone at high risk (subjects residing around an index case), rather than rely on RDT results, which have been shown to miss infections. In a low transmission setting such as Namibia, only a small proportion of the populations is at high risk of infection, therefore, only a small number of people need to be targeted (perhaps 20-50 people). Additional indoor residual spraying (IRS) targeted to homes in high risk locations can also be implemented.

rfMDA is a promising strategy, but evidence does not yet exist to prove its efficacy in Africa. Questions remain about where to target rfMDA, what drugs to use, and whether drugs should be used alone or in combination with additional vector control. For rfMDA to be most successful, it is necessary to kill parasites in the human as well as the vector population of the target area. However, one challenge of pre-transmission season IRS is that it is difficult to predict where future infections will occur. A reactive approach, in conjunction with the pre-transmission approach, will ensure coverage of effective vector control in the highest risk areas. Further, if there is unknown resistance to the insecticide used during pre-transmission season, the subsequent reactive use of a different, and presumably effective insecticide, will provide better protection.

In this study the investigators will utilise a cluster randomized controlled study design to evaluate rfMDA in response to a passively identified index case and compare it to RACD. The investigators will study each intervention (rfMDA, RACD) both with and without additional focal insecticide spraying.

56 enumeration areas (EAs) within catchment areas of 11 study health facilities will be randomized to one of four intervention arms:

1. RACD only
2. RACD with RAVC
3. rfMDA only
4. rfMDA with RAVC

A rapid reporting surveillance system will capture confirmed, passively identified cases at all study health facilities, and those cases will trigger an intervention by the study team if located in one of the study EAs.

ELIGIBILITY:
Inclusion Criteria:

1. Index Case Investigation Inclusion Criteria:

   * Malaria infection (either locally transmitted or imported) detected at a health facility via passive surveillance, and
   * Resides in a study Enumeration Area (EA), and
   * Provides informed consent
2. RACD Intervention Inclusion Criteria:

   * Provides informed consent, and
   * Index case resides in study EA, and
   * All non-index cases that reside or spent at least one night in the Target Area in the past 4 weeks, and
   * Residents of the six houses closest to the index case, and
   * If 25 people are not enrolled in the study at the first six houses, plus the index case household, after the second visit then additional houses can be approached on the third visit.
3. rfMDA Intervention Inclusion Criteria:

   * Provides informed consent, and
   * Index case resides in study EA, and
   * All non-index cases that reside or spent at least one night in the Target Area in the past 4 weeks, and
   * Residents of the six houses closest to the index case, and
   * If 25 people are not enrolled in the study at the first six houses, plus the index case household, after the second visit then additional houses can be approached on the third visit.
4. Artemether/Lumefantrine (A-L) (combination medication) Inclusion Criteria:

   * Consent to take A-L medication
   * Does not meet A-L Exclusion Criteria under item #4 below
5. Pill count Inclusion Criteria:

   * Provides consent, and
   * People who receive any number of RACD or rfMDA drug dose(s)
6. Reactive Vector Control Inclusion Criteria:

   * Informed consent provided by head of household or person in otherwise in charge of household, and
   * Index case resides in study EA, and
   * Index household and 6 non-index households closest to index household
7. Endline Survey, Individual, Inclusion Criteria:

   * Provides informed consent, and
   * Resides or spent at least 1 night in the EA in the preceding 4 weeks
8. Acceptability Assessment: Individual Interviews with study participants, Inclusion Criteria:

   * Provides informed consent, and
   * Resident of index household or of neighbouring households
9. Acceptability Assessment: Individual Interviews with key stakeholders, Inclusion Criteria:

   * In leadership position within Zambezi region, and
   * Provides informed consent
10. Acceptability Assessment: Individual Interview with refusers, Inclusion Criteria:

    * Refused to participate in rfMDA, RACD, and/or RAVC, and
    * Provides informed consent to take part in the anonymous survey
11. Acceptability Assessment: Focus group discussions with study participants, Inclusion Criteria:

    * Provides informed consent, and
    * Was eligible to be enrolled in the study in participant's Target Area, and
    * Either took part in RACD or rfMDA intervention (+/- RAVC), OR refused these interventions

Exclusion Criteria:

1. Index Case Investigation Exclusion Criteria:

   * Malaria infection identified through active case detection
   * Refusal to participate
2. RACD Intervention Exclusion Criteria:

   * Index case does not reside in study EA, or
   * Refusal to participate in RACD, or
   * Household received the intervention in the previous 5 weeks, or
   * Household > 500 m from the index case, or
   * Severe or complicated malaria as assessed by study nurse (this will lead to referral for further evaluation at health facility but not enrolment in study)
3. rfMDA Intervention Exclusion Criteria:

   * Index case does not reside in study EA, or
   * Refusal to participate in rfMDA, or
   * Household received the intervention in the previous 5 weeks, or
   * Household > 500 m from the index case, or
   * Severe or complicated malaria as assessed by study nurse (this will lead to referral for further evaluation at health facility but not enrolment in study)
4. Artemether/Lumefantrine (combination medication) Exclusion Criteria:

   * Pregnancy in first trimester, or
   * Previous regular menstruation, with no menstruation for most recent 4 weeks, or
   * Weight < 5 kg*, or
   * Severe malaria, or
   * Known allergy to A-L, or
   * Refusal of the offered A-L

     * Note regarding A-L weight exclusion: Because of the pre-set required field at the top of the Eligibility section of this Application, the investigators have indicated a 6 month minimum age limit, primarily to note to the reader that there will be a lower age limit to infants enrolled. Yet during the actual conduct of this trial the investigators will utilize 5 kg weight as the cutoff, rather than using age. A lower weight cutoff of 5 kg is in accordance with A-L's manufacturer (Novartis)'s guidance on supporting pediatric data.
5. Pill count Exclusion Criteria:

   * Refusal to participate in pill count, or
   * Individuals who did not receive any drug doses through RACD or rfMDA
6. Reactive Vector Control Exclusion Criteria:

   * Refusal by head of household to participate in RAVC, or
   * Already received RAVC during current transmission season, or
   * Household is > 500 m from index case household (note: refusal to participate in RACD or rfMDA is not an exclusion criterion for RAVC)
7. Endline Survey, Individual, Exclusion Criteria:

   • Refusal to participate in Endline Survey (note: lack of participation in rfMDA or RACD is not an exclusion criterion)
8. Acceptability Assessment: Individual Interviews with study participants, Exclusion Criteria:

   * Refusal to participate in Acceptability Assessment, or
   * Speaks language not understood or able to be translated, or
   * Key stakeholder [see below]
   * Age < 15 years
9. Acceptability Assessment: Individual Interviews with key stakeholders, Exclusion Criteria:

   * Refusal to participate in Acceptability Assessment, or
   * Speaks language not understood or able to be translated, or
   * Not in leadership position
10. Acceptability Assessment: Individual Interview with refusers, Exclusion Criteria:

    * Refusal to participate in Acceptability Assessment, or
    * Speaks language not understood or able to be translated, or
    * Age < 15 years
11. Acceptability Assessment: Focus group discussions with study participants, Exclusion Criteria:

    * Refusal to participate in Acceptability Assessment, or
    * Speaks language not understood or able to be translated, or
    * Key stakeholder or in another leadership position, or
    * Age < 15 years

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9845 (Actual)
Dates: Start 2016-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Incidence | Up to 12 months
  Incidence of confirmed, passively identified malaria cases

SECONDARY OUTCOMES:
All-age infection prevalence | Up to 12 months
  The investigators will determine all-age infection prevalence using loop-mediated isothermal amplification (LAMP) during the cross-sectional household survey. This survey will be administered to a sample of residents of all intervention Enumeration Areas in the Study Area at study conclusion.
All-age seroprevalence | Up to 12 months
  The investigators will determine all-age seroprevalence using ELISA during the cross-sectional household survey. This survey will be administered to a sample of residents of all intervention EAs in the Study Area at study conclusion.
Feasibility of attaining coverage | Up to 12 months
  The investigators will compare coverage of each intervention package and determine the feasibility of reaching 80% coverage for each intervention package. For RACD intervention, this equates to the proportion of the population living in the Target Area that receives a finger prick to test for malaria. For TPE intervention, coverage equates to the proportion that receive an initial dose of antimalarial drug (intention to treat analysis). For RAVC intervention, coverage is defined as the proportion of houses in the Target Area that receive reactive Indoor Residual Spraying (IRS).
Safety: Serious adverse events (SAEs) | Up to 12 months
  The investigators will compare the count of serious adverse events (SAEs) relative to the total number of participants receiving an Intervention, across interventions.
Acceptability | Up to 12 months
  Using focus group discussions (FGDs), the investigators will ask two questions: "Was this intervention acceptable to [participant]?" and "Would [participant] participate in this intervention again if given the opportunity?". The investigators will compare the % of "yes" responses to each of these questions, in the TPE versus the RACD arms.
Refusal rates | Up to 12 months
  Refusal rates for each intervention
Cost of intervention | Up to 12 months
  The investigators will collect detailed expenditure data on costs of delivery of the TPE and RACD interventions. Calculations will include costs for all consumables, as well as staff time, which will be prospectively collected every 10th TPE or RACD event. The investigators will compare TPE versus RACD in terms of cost per intervention event as well as cost per population intervened upon.
Medication adherence | Up to 12 months
  The investigators will measure medication adherence in both TPE and RACD by scheduled pill counts in a random subset of subjects receiving each of those interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hsiang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of Namibia Multidisciplinary Research Centre, Windhoek, Namibia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bousema T, Griffin JT, Sauerwein RW, Smith DL, Churcher TS, Takken W, Ghani A, Drakeley C, Gosling R. Hitting hotspots: spatial targeting of malaria for control and elimination. PLoS Med. 2012 Jan;9(1):e1001165. doi: 10.1371/journal.pmed.1001165. Epub 2012 Jan 31. PMID 22303287
- [Background] Moonen B, Cohen JM, Snow RW, Slutsker L, Drakeley C, Smith DL, Abeyasinghe RR, Rodriguez MH, Maharaj R, Tanner M, Targett G. Operational strategies to achieve and maintain malaria elimination. Lancet. 2010 Nov 6;376(9752):1592-603. doi: 10.1016/S0140-6736(10)61269-X. Epub 2010 Oct 28. PMID 21035841
- [Background] Carter R, Mendis KN, Roberts D. Spatial targeting of interventions against malaria. Bull World Health Organ. 2000;78(12):1401-11. Epub 2003 Nov 17. PMID 11196487
- [Background] Hsiang MS, Hwang J, Kunene S, Drakeley C, Kandula D, Novotny J, Parizo J, Jensen T, Tong M, Kemere J, Dlamini S, Moonen B, Angov E, Dutta S, Ockenhouse C, Dorsey G, Greenhouse B. Surveillance for malaria elimination in Swaziland: a national cross-sectional study using pooled PCR and serology. PLoS One. 2012;7(1):e29550. doi: 10.1371/journal.pone.0029550. Epub 2012 Jan 6. PMID 22238621
- [Background] Sturrock HJ, Novotny JM, Kunene S, Dlamini S, Zulu Z, Cohen JM, Hsiang MS, Greenhouse B, Gosling RD. Reactive case detection for malaria elimination: real-life experience from an ongoing program in Swaziland. PLoS One. 2013 May 20;8(5):e63830. doi: 10.1371/journal.pone.0063830. Print 2013. PMID 23700437
- [Background] Hsiang MS, Hwang J, Tao AR, Liu Y, Bennett A, Shanks GD, Cao J, Kachur SP, Feachem RG, Gosling RD, Gao Q. Mass drug administration for the control and elimination of Plasmodium vivax malaria: an ecological study from Jiangsu province, China. Malar J. 2013 Nov 1;12:383. doi: 10.1186/1475-2875-12-383. PMID 24175930
- [Background] Oxborough RM, Kitau J, Jones R, Feston E, Matowo J, Mosha FW, Rowland MW. Long-lasting control of Anopheles arabiensis by a single spray application of micro-encapsulated pirimiphos-methyl (Actellic(R) 300 CS). Malar J. 2014 Jan 29;13:37. doi: 10.1186/1475-2875-13-37. PMID 24476070
- [Background] White NJ. Intermittent presumptive treatment for malaria. PLoS Med. 2005 Jan;2(1):e3. doi: 10.1371/journal.pmed.0020003. PMID 15696210
- [Background] Katrak S, Gasasira A, Arinaitwe E, Kakuru A, Wanzira H, Bigira V, Sandison TG, Homsy J, Tappero JW, Kamya MR, Dorsey G. Safety and tolerability of artemether-lumefantrine versus dihydroartemisinin-piperaquine for malaria in young HIV-infected and uninfected children. Malar J. 2009 Nov 30;8:272. doi: 10.1186/1475-2875-8-272. PMID 19948038
- [Background] Banek K, Lalani M, Staedke SG, Chandramohan D. Adherence to artemisinin-based combination therapy for the treatment of malaria: a systematic review of the evidence. Malar J. 2014 Jan 6;13:7. doi: 10.1186/1475-2875-13-7. PMID 24386988
- [Derived] Ntuku H, Smith-Gueye C, Scott V, Njau J, Whittemore B, Zelman B, Tambo M, Prach LM, Wu L, Schrubbe L, Kang Dufour MS, Mwilima A, Uusiku P, Sturrock H, Bennett A, Smith J, Kleinschmidt I, Mumbengegwi D, Gosling R, Hsiang M. Cost and cost effectiveness of reactive case detection (RACD), reactive focal mass drug administration (rfMDA) and reactive focal vector control (RAVC) to reduce malaria in the low endemic setting of Namibia: an analysis alongside a 2x2 factorial design cluster randomised controlled trial. BMJ Open. 2022 Jun 23;12(6):e049050. doi: 10.1136/bmjopen-2021-049050. PMID 35738650
- [Derived] Hsiang MS, Ntuku H, Roberts KW, Dufour MK, Whittemore B, Tambo M, McCreesh P, Medzihradsky OF, Prach LM, Siloka G, Siame N, Gueye CS, Schrubbe L, Wu L, Scott V, Tessema S, Greenhouse B, Erlank E, Koekemoer LL, Sturrock HJW, Mwilima A, Katokele S, Uusiku P, Bennett A, Smith JL, Kleinschmidt I, Mumbengegwi D, Gosling R. Effectiveness of reactive focal mass drug administration and reactive focal vector control to reduce malaria transmission in the low malaria-endemic setting of Namibia: a cluster-randomised controlled, open-label, two-by-two factorial design trial. Lancet. 2020 Apr 25;395(10233):1361-1373. doi: 10.1016/S0140-6736(20)30470-0. PMID 32334702
- [Derived] Medzihradsky OF, Kleinschmidt I, Mumbengegwi D, Roberts KW, McCreesh P, Dufour MK, Uusiku P, Katokele S, Bennett A, Smith J, Sturrock H, Prach LM, Ntuku H, Tambo M, Didier B, Greenhouse B, Gani Z, Aerts A, Gosling R, Hsiang MS. Study protocol for a cluster randomised controlled factorial design trial to assess the effectiveness and feasibility of reactive focal mass drug administration and vector control to reduce malaria transmission in the low endemic setting of Namibia. BMJ Open. 2018 Jan 27;8(1):e019294. doi: 10.1136/bmjopen-2017-019294. PMID 29374672

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT02610400/Prot_SAP_001.pdf